CLINICAL TRIAL: NCT01576900
Title: The Effect of Combined Systematized Behavioural Modification Education Program (SyBeMeP) With DDAVP in Patients With Nocturia
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Seung-June Oh, Professor, Seoul National University Hospital
Other Study IDs: Nocturia-SBMP
Record Dates: First submitted 2012-02-13; First posted 2012-04-13 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Nocturia
Keywords: behavior therapy; nocturia; polyuria
MeSH Terms: conditions — Nocturia; Polyuria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Desmopressin monotherapy: Control group: Desmopressin (Minirin Tablet 0.1-0.4mg/day) + simple instruction
- Combination group: Study group: Desmopressin (Minirin Tablet 0.1-0.4mg/day) + SyBeMeP
  * Patients will be randomized and assigned to each group at the ratio of 1:1.
  Interventions: Behavioral: SyBeMeP (Systemized Behavioural Modification education Program)

INTERVENTIONS:
Behavioral: SyBeMeP (Systemized Behavioural Modification education Program) — * Standard video material will be developed to minimize variation of outcomes caused by differences in contents at each trial site.
  * Video material will be self-study program for PC with running time around 20 minutes. Contents will cover pathophysiology, diagnosis and treatment process, and be easy to understand for everyone with variety of examples. In treatment part, it will describe general principles of behavioural therapy (Adjustment of timing of fluid intake, Reducing alcohol and caffeine, Improving sleep hygiene including moderate exercise, room temperature, noise and lighting. if necessary, compressive stocking, late afternoon nap and leg elevation would be added)
  * During trial, patients will watch SYBeMeP at a specially prepared separate room with computer.
  * After watching the video, check-list on take-home message will be recorded by patients at the site to confirm patients' awareness after education.
  Groups: Combination group

SUMMARY:
In patients with nocturia, combinational treatment of DDAVP and SyBeMeP might show better outcomes.

Systemic video instruction might prove to be beneficial by helping patients have better understanding on treatment and replacing healthcare personnel.

DETAILED DESCRIPTION:
One of main reason of nocturia is known as nocturnal polyuria. For the treatment of nocturia caused by overactive bladder, the combined therapy of anticholinergics plus behavioural modification has been established as the first line therapy. However, nocturia mainly comes from polyuria has been treated with desmopressin pharmacotherapy and the effect of behaviour modification education has not yet evaluated. Therefore, in this study, short term synergistic effect of combinational treatment of desmopressin and SyBeMeP (Systemized Behavioral Modification education Program) comparing desmopressin monotherpy will be evaluated in patients with nocturia.

Control group: Desmopressin (Minirin Tablet 0.1-0.4mg/day) + simple instruction Study group: Desmopressin (Minirin Tablet 0.1-0.4mg/day) + SyBeMeP. Patients will be randomized and assigned to each group at the ratio of 1:1. At screening visit, flowmetry and residual urine measurement, Complete Blood Count (CBC), atypical diabetes mellitus (ADM), electrolytes, urinalysis micro, urine concentration, and demographic examination will be done. Voiding diary will be distributed. At 2nd visit, patients will be randomized and each treatment will be initiated. IPSS, ICIQ-nocturia, and PPTB will be completed. Voiding diary will be distributed. At 3rd visit (2 weeks after from 2nd visit): IPSS, ICIQ-nocturia, and PPTB will be completed. Assess the treatment outcome including voiding diary analysis.

ELIGIBILITY:
Inclusion Criteria:

* A patient with nocturia, who visited department of urology as outpatient
* Have not been treated with desmopressin for at least 6 months before

Exclusion Criteria:

* Sleep disorder,
* history of medication for voiding,
* diabetes insipidus,
* diabetes mellitus,
* cardiovascular disease,
* voiding difficulties (including residual urine of more than 100ml),
* small bladder capacity,
* overactive bladder,
* illiteracy,
* psychiatric disorder and having no intention to be enrolled by written agreement

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean patients with nocturia regardless of age and gender
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2012-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Decrease in urinary frequency (No. of nocturia) | baseline, 2 week, 1 month, and 3 months

SECONDARY OUTCOMES:
Voiding diary indices | baseline, 2 weeks, 1 month and 3 months
IPSS | baseline, 2 weeks, 1 month and 3 months
ICIQ-nocturia | baseline, 2 weeks, 1 month and 3 months
patient's perception of bladder condition (PPTB) | baseline, 2 weeks, 1 month and 3 months
patient's satisfaction on the education | baseline, 2 weeks, 1 month and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sung Yong Cho, M.D.,Ph.D., Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Cho SY, Lee SL, Kim IS, Koo DH, Kim HJ, Oh SJ. Short-term effects of systematized behavioral modification program for nocturia: a prospective study. Neurourol Urodyn. 2012 Jan;31(1):64-8. doi: 10.1002/nau.21186. Epub 2011 Aug 8. PMID 21826726